CLINICAL TRIAL: NCT04843774
Title: Vaccine-generated Immunity in Ocrelizumab-treated Patients: Longitudinal Assessments (VIOLA)
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 21-00206
Record Dates: First submitted 2021-04-09; First posted 2021-04-14 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
Keywords: SARS-CoV-2 Vaccine; Ocrelizumab
MeSH Terms: conditions — Multiple Sclerosis | interventions — CVnCoV COVID-19 vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patients will have 5 blood draws in-person
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- COVID-negative Multiple Sclerosis patients treated with ocrelizumab
  Interventions: Drug: SARS-COV-2 mRNA Vaccine

INTERVENTIONS:
Drug: SARS-COV-2 mRNA Vaccine — Pfizer-BioNTech and Moderna messenger RNA (mRNA)-platform vaccines developed against SARS-CoV-2 virus will be given as standard of care (SOC)

SUMMARY:
Severe acute respiratory coronavirus 2 (SARS-CoV-2) is a novel coronavirus and the causative agent of COVID 19 disease, whose presentation symptoms range from asymptomatic infection to mild flu-like symptoms to multi system failure and death, resulting in significant morbidity and mortality worldwide. Novel vaccines against the SARS-CoV-2 virus have very recently been developed; however, the effectiveness, immune response, and short- or long-term safety of these vaccines have not been tested in immunocompromised patients on anti-CD-20 therapy for multiple sclerosis (MS) or for other disorders.

This study will examine the immune response of the Pfizer-BioNTech and Moderna messenger RNA (mRNA)-platform vaccines developed against SARS-CoV-2 virus given as standard of care (SOC) in MS patients on ocrelizumab.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent and understand and agree to be compliant with the study protocol
* Age 18 to 65 years at time of signing the ICF
* For women of childbearing potential: agreement to avoid in-vitro fertilization or remain abstinent (refrain from heterosexual intercourse) or use acceptable contraceptive methods during the treatment period and for 6 months after the final dose of ocrelizumab

  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). The definition of childbearing potential may be adapted for alignment with local guidelines or requirements.
  * The following are acceptable contraceptive methods (as defined by the guidelines): progesterone-only hormonal contraception, where inhibition of ovulation is not the primary mode of action; male or female condom with or without spermicide; and cap, diaphragm, or sponge with spermicide. More effective contraceptive methods (e.g., bilateral tubal ligation; male sterilization; copper intrauterine devices) may be used, but are not required.
* Diagnosis of RMS, PPMS, SPMS currently on ocrelizumab therapy
* Patients on ocrelizumab as SOC with the last dose received within 6 months prior to first vaccine
* EDSS <= 6.5
* Able to comply with study procedures based on the assessment of the Investigator
* Healthy adults or adults with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.

Exclusion Criteria:

* MS related

  * Clinical MS relapse as defined by the treating physician, documented within the last 3 months prior to vaccine
  * Is acutely ill or febrile 72 hours prior to or at screening. Fever is defined as a body temperature >=38.0C/100.4F. Participants meeting this criterion may be rescheduled within the relevant window periods. Febrile participants with minor illnesses can be enrolled at the discretion of the investigator.
* Is pregnant or breastfeeding; women of childbearing potential must have a negative serum or urine pregnancy test result within 14 days prior to study enrollment
* Known history of SARS-CoV-2 infection as defined by:

  1. Meeting CDC Clinical Case Definition Criteria (CDC, 2020) in which at least two core symptoms below are present:

     * New continuous cough,
     * Temperature >= 37.8C,
     * Loss of, or change in, normal sense of smell (anosmia) or taste (ageusia) in the absence of alternative explanation,
     * Additional features such as influenza-like illness, clinical or radiological evidence of pneumonia, or acute worsening of underlying respiratory illness, or fever without another cause, AND
  2. Objective evidence that supports COVID 19 diagnosis, such as detection of SARS-CoV-2 specific antibody in serum, plasma, or whole blood; radiographic evidence of pneumonia or acute respiratory distress syndrome.
* Prior mRNA vaccine for COVID 19
* History of a delayed second dose of vaccine >= 14 days from recommended dosing
* Prior administration of an investigational coronavirus (SARS CoV, MERS CoV) vaccine or current/planned simultaneous participation in another interventional study to prevent or treat COVID 19
* Demonstrated inability to comply with the study procedures
* Known or suspected allergy or history of anaphylaxis, urticaria, or other significant adverse reaction to the vaccine or its excipients
* Bleeding disorder considered a contraindication to intramuscular injection or phlebotomy
* Has received or plans to receive a non-study vaccine within 28 days prior to or after any dose of COVID vaccine (except for seasonal influenza vaccine, which is not permitted within 14 days before or after any dose of COVID vaccine)
* Has participated in an interventional clinical study within 28 days prior to the day of enrollment
* Immunosuppressive or immunodeficient state, asplenia, recurrent severe infections (HIV-positive participants with CD4 count >=350 cells/mm^3 and an undetectable HIV viral load within the past year [low-level variations from 50 to 500 viral copies that do not lead to changes in antiretroviral therapy are permitted])
* Has received systemic steroids or other immunosuppressants other than those required as ocrelizumab pre-medication for >14 days in total within 6 months prior to screening (for corticosteroids >=20 mg/day of prednisone equivalent)
* Has received high-dose intravenous (IV) or oral steroids within 30 days of screening; IVIG or PLEX within 3 months of screening
* Has received systemic immunoglobulins or blood products within 3 months prior to the day of screening
* Patients cannot receive other COVID 19 vaccine products outside this study during the study period
* Infection related

  - Known active bacterial, viral, fungal, mycobacterial infection, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infection of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks prior to baseline visit or oral antibiotics within 2 weeks prior to baseline visit
* Cancer Related

  - History of cancer, including solid tumors and hematological malignancies (except basal cell, in situ squamous cell carcinomas of the skin, and in situ carcinoma of the cervix or the uterus that have been excised and resolved with documented clean margins on pathology)
* Other medical conditions

  * History of or currently active primary or secondary immunodeficiency
  * History of active alcohol or other drug abuse
  * Any concomitant, non-MS disease that may require chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
  * Significant, uncontrolled disease, as defined by AMA guidelines or similar, such as cardiovascular (including congestive heart failure - NYHA Grade 3 or 4, cardiac arrhythmia), uncontrolled hypertension, pulmonary (including chronic obstructive pulmonary disease), renal, hepatic, endocrine (including uncontrolled diabetes mellitus), and gastrointestinal
  * Known presence or history of other neurologic disorders, including but not limited to, the following:

    * Neuromyelitis optica spectrum disorders (NMOSD)
    * Severe, clinically significant brain or spinal cord trauma (e.g., cerebral contusion, spinal cord compression)
    * Psychosis not yet controlled by a treatment
* Prior DMT for MS

  * Previous treatment with alemtuzemab, cyclophosphamide, mitoxantrone, azathioprine, mycophenolate mofetil, cyclosporine, methotrexate, total body irradiation, or bone marrow transplantation
  * Treatment with another anti-CD 20 depleting agent within 6 months
* Laboratory - Certain laboratory abnormalities or findings at screening, including the following:

  * IgG <300, or patients trending toward <300 based on previous labs/trajectory (PI discretion) at time of screening labs
  * Absolute lymphocyte count <750/mm3 at time of screening labs
  * Absolute neutrophil count <1000/mm3 at time of screening labs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: COVID-negative Multiple Sclerosis patients treated with ocrelizumab
Sampling Method: Non-Probability Sample
Enrollment: 64 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Anti-SARS-CoV-2 S Titer Levels | Baseline, Pre-First Vaccine Dose
Anti-SARS-CoV-2 S Titer Levels | Week 4, Post-Last Dose of Vaccine
Anti-SARS-CoV-2 S Titer Levels | Week 12, Post-Last Dose of Vaccine
Number of participants with a fold rise of serum anti-SARS-CoV-2 S titers | Baseline, Pre-First Vaccine Dose
  This outcome measure will be reported for participants with a fold rise >=2, >=3, and >=4 of serum anti-SARS-CoV-2 S titers
Number of participants with a fold rise of serum anti-SARS-CoV-2 S titers | Week 4, Post-Last Dose of Vaccine
  This outcome measure will be reported for participants with a fold rise >=2, >=3, and >=4 of serum anti-SARS-CoV-2 S titers
Number of participants with a fold rise of serum anti-SARS-CoV-2 S titers | Week 12, Post-Last Dose of Vaccine
  This outcome measure will be reported for participants with a fold rise >=2, >=3, and >=4 of serum anti-SARS-CoV-2 S titers
T-Cell Response | Baseline, Pre-First Vaccine Dose
  T-cell response will be measured by ELISpot assay
T-Cell Response | Week 4, Post-Last Dose of Vaccine
  T-cell response will be measured by ELISpot assay
T-Cell Response | Week 12, Post-Last Dose of Vaccine
  T-cell response will be measured by ELISpot assay

SECONDARY OUTCOMES:
SARS-CoV-2 anti-S1 and anti-Receptor Binding Domain (RBD) binding antibody levels | Week 4, Post-Last Dose of Vaccine
SARS-CoV-2 anti-S1 and anti-Receptor Binding Domain (RBD) binding antibody levels | Week 12, Post-Last Dose of Vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Ilya Kister, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - University of Colorado, Denver (UCD), Denver, Colorado
  - NYU Langone Health Multiple Sclerosis Comprehensive Care Center (NYULH MSCCC), New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Curtin R, Velmurugu Y, Dibba F, Hao Y, Sreenivasaiah C, Khodadadi-Jamayran A, Nyovanie S, Kim A, Samanovic ML, Mulligan M, Priest J, Cabatingan M, Winger RC, Patskovsky Y, Kister I, Silverman GJ, Krogsgaard M. Persistent Classical and Atypical Memory B Cells Underlie Heterogeneous Vaccine Responses in Ocrelizumab-Treated Multiple Sclerosis. bioRxiv [Preprint]. 2025 Nov 4:2025.11.03.686372. doi: 10.1101/2025.11.03.686372. PMID 41279857